CLINICAL TRIAL: NCT06923332
Title: A Randomized, Crossover Trial to Assess the Effects of Short-term Diets With and Without Inulin on Energy Expenditure in Adults
Brief Title: A Trial to Assess the Effects of Diets With and Without Inulin on Energy Expenditure in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2430
Record Dates: First submitted 2025-04-02; First posted 2025-04-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Overweight or Obese Adults
MeSH Terms: conditions — Overweight | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin - high fiber (Experimental)
  Interventions: Other: High Fiber bar with Inulin
- Control - Low Fiber (Active Comparator)
  Interventions: Other: Low fiber bar - no inulin

INTERVENTIONS:
Other: High Fiber bar with Inulin — Bar with inulin - high fiber
  Arms: Inulin - high fiber
Other: Low fiber bar - no inulin — Bar without inulin - low fiber
  Arms: Control - Low Fiber

SUMMARY:
The objective of this trial is to assess the effects of a 7-day diet containing inulin vs. a control diet on energy expenditure in adults with overweight/obesity or normal weight.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years of age, inclusive. There will be approximately equal numbers of men and women.
2. Individual has BMI of 18.5 to 24.9 kg/m2 or 27.0 to 34.9 kg/m2, inclusive.
3. Premenopausal women that are not using hormonal contraceptives must have a history of regular menstrual cycles (21-35 days per cycle) for at least 3 months prior to visit 1.
4. Individual is judged by the Investigator to be in generally good health on the basis of medical history and screening measurements.
5. Individual is willing and able to undergo the scheduled study procedures.
6. Individual understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Individual has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
2. Individual has a clinically significant medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results. Health conditions may include history or presence of clinically important GI, cardiac, renal, hepatic, endocrine (i.e., diabetes), pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator. Clinically important GI conditions included but are not limited to: inflammatory bowel disease, irritable bowel syndrome, gastroparesis, clinically important lactose intolerance.
3. Individual habitually consumes >8 g fiber per 1000 kcal per day. A 14-day washout prior to the first test and throughout the study period is permitted.
4. Individual habitually consumes fiber supplements. A 14-day washout prior to the first test and throughout the study period is permitted.
5. Use of tobacco/nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of visit 1.
6. Use of hemp/marijuana products within 12 months of visit 1. Occasional use (e.g., once or twice a month) within 12 months of visit 1 is allowed but requires at least a 14-day washout prior to visit 1 and the participant must be willing to refrain from use during the study.
7. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.
8. Individual has used an alpha-blocker, beta-blocker, or high-dose diuretic within 30 days of visit 1. Unstable use (initiation or change in dose) within 30 days of visit 1 of other antihypertensive medications is also exclusionary.
9. Unstable use (initiation or change in dose) within 30 days of visit 1 of thyroid hormone replacement medications.
10. Unstable use (initiation or change in dose) within 30 days of visit 1 of sex hormones. Multiphasic hormonal contraceptives in which the amount of sex hormone in the active pill varies by week (i.e., biphasic, triphasic, quadriphasic) are considered unstable doses of sex hormones and are exclusionary.
11. Use of medications or supplements that may influence carbohydrate or fat metabolism, including but not limited to hypoglycemic medications and systemic (intravenous, intramuscular, or oral) or ≥1500 µg/day (topical, inhaled, intranasal, or dermal) corticosteroids within 30 days of visit 1.
12. Use of any weight loss medication within 90 days of visit 1.
13. Use of medications or supplements that may influence heart rate, including but not limited to stimulant medications (e.g., amphetamines, methylphenidates, etc.) within 30 days of visit 1.
14. Use of digestive enzymes, prebiotics, probiotics, and/or postbiotics within 14 days of the first test visit and throughout the study period.
15. Individual has a history of cancer in the prior 5 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
16. Individual has had a weight change of ± 4.5 kg (10 lb.) in the previous 3 months.
17. Individual has extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian).
18. Individual is actively following a weight loss diet (even if maintaining body weight).
19. Individual has a history of bariatric surgery or is actively attempting to lose or gain body weight.
20. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
21. History of any major trauma or major surgical event within 2 months of visit 1.
22. Individual has signs or symptoms of an active infection of clinical significance or has taken antibiotics within 5 days prior to any visit (washout is permitted for re-scheduling of the clinic visit).
23. Individual has an allergy, sensitivity or intolerance to any components of the study product or study meals.
24. Individual is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
25. Individual has been exposed to any non-registered drug product within 30 days prior to screening.
26. Individual has a current or recent history (within 12 months prior to screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz. beer, 5 oz. wine, or 1.5 oz. hard liquor).
27. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Measured in kcal/day

SECONDARY OUTCOMES:
Diet Induced Thermogenesis | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the full test period
Diet Induced Thermogenesis | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the breakfast period
Diet Induced Thermogenesis | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the lunch period
Postprandial carbohydrate oxidation rate | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the full test period
Postprandial carbohydrate oxidation rate | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the breakfast period
Postprandial carbohydrate oxidation rate | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the lunch period
Postprandial fat oxidation rate | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the full test period
Postprandial fat oxidation rate | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the breakfast period
Postprandial fat oxidation rate | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the lunch period
Postprandial respiratory exchange ration (RER) | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the full test period
Postprandial respiratory exchange ration (RER) | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the breakfast period
Postprandial respiratory exchange ration (RER) | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Assessed as the AUC and niAUC during the lunch period
Fasting Carbohydrate Oxidation | pre-consumption
  Assessed from pre-consumption
Fasting Fat Oxidation | pre-consumption
  Assessed from pre-consumption
Fasting RER | pre-consumption
  Assessed from pre-consumption
Fat Mass | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Measured using the Styku body scanner.
Fat-Free Mass | Measured on days 7 and 21 where days 1 and 15 are the first day of study product intake for each treatment. Day 7 to 14 is the washout period.
  Calculated by subtracting fat mass from body mass.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research and Consulting LLC
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No